CLINICAL TRIAL: NCT06544551
Title: Efficacy and Safety Study of Peginterferon Alfacon-2 to Treat Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Kawin Technology Share-Holding Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Junqi Niu, Principal Investigator, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kawin-2021-001
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peginterferon Alfacon-2 treated patients (Experimental)
  Interventions: Drug: Peginterferon Alfacon-2
- Peginterferon Alfacon-2 placebo treated patients (Placebo Comparator)
  Interventions: Drug: Peginterferon Alfacon-2 placebo

INTERVENTIONS:
Drug: Peginterferon Alfacon-2 — Peginterferon Alfacon-2 injection will be weekly subcutaneous injected for 48 weeks. Tenofovir alafenamide Fumarate Tablets(TAF) will be take orally for at least 48 weeks, not more than 72 weeks. Peg-interferon Alfacon-2 and TAF will discontinue when HBsAg levels is less than 0.05 IU/mL and HBV DNA is below 10 IU/mL during 48-72 weeks.
  Arms: Peginterferon Alfacon-2 treated patients
Drug: Peginterferon Alfacon-2 placebo — Peginterferon Alfacon-2 placebo injection will be weekly subcutaneous injected for 48 weeks. Tenofovir alafenamide Fumarate Tablets(TAF) will be take orally for at least 48 weeks, not more than 72 weeks. Peg-interferon Alfacon-2 and TAF will discontinue when HBsAg levels is less than 0.05 IU/mL and HBV DNA is below 10 IU/mL during 48-72 weeks.
  Arms: Peginterferon Alfacon-2 placebo treated patients

SUMMARY:
Current clinical practices has shown promising prospects of the therapy strategy of interferon combined with nucleos(t)ides in patients with chronic hepatitis B, but the safety and efficacy has not been fully studied. This study is aimed to exploit the safety and efficacy of the study drug, Peginterferon Alfacon-2 injection, with nucleos(t)ide (NAs), Tenofovir alafenamide Fumarate Tablets (TAF), in the patients with hepatitis B virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years (including 18 and 60), no gender limit.
* BMI between 18 and 30 kg/m2 (including 18 and 30).
* For treatment naive patients: Did not receive standard anti-HBV treatment within 6 months prior to screening (Including interferon, NAs, and other anti-HBV drugs).
* For NAs treated patients: Who should have continuously taken NAs for at least 9 months prior to screening, and are currently receiving the NAs.
* HBsAg positive for at least 6 months and HBsAg between 10 and 1000 IU/mL (excluding 10 and 1000).
* HBsAb and HBeAg both are negative at screening.
* For treatment naive patients: HBV DNA < 2×10^3 IU/mL at screening.
* For NAs treated patients: HBV DNA < 100 IU/mL at screening.
* For treatment naive patients: ALT ≤ 5ULN at screening.
* For NAs treated patients: ALT ≤ 2ULN at screening.
* Liver stiffness measurement <8.0 kPa at screening.
* Pregnancy test of female of childbearing must be negative at screening, and the subjects (male and female) should take effective contraceptive measures during the whole study period.
* Understand and sign the informed consent form voluntarily.

Exclusion Criteria:

* For NAs treated patients: who have received standard treatment of interferon products within 6 months prior to screening.
* Systemic therapy with potent immunomodulatory agents such as adrenocorticotropic hormone, thymosin α1, etc more than two weeks within past 6 months, not including corticosteroid nasal sprays, inhaled steroids and / or topical steroids.
* Co-infected with Hepatitis A, Hepatitis C, Hepatitis D, Hepatitis E, or HIV.
* Evidence of liver compensation, including previous liver biopsy, imaging examination or clinical manifestations.
* Evidences of hepatic decompensation, including but not limited to serum total bilirubin> 2 times the upper limit of normal (ULN); serum albumin <35g/L; prothrombin activity (PTA) <60%; ascites, upper gastrointestinal bleeding and hepatic encephalopathy; Child-Pugh score B/C grade.
* Evidence of hepatocellular carcinoma, or AFP>>50 ng/mL, or imaging examination revealed suspicious nodules in the liver.
* Liver diseases from other causes, including alcoholic liver disease, non-alcoholic steatohepatitis, drug-induced hepatitis, autoimmune hepatitis (antinuclear antibody titer higher than 1:100), hepatolenticular degeneration (Wilson's disease) and hemochromatosis, etc.
* White blood cell count <3×10^9/L; neutrophil count<1.5×10^9/L; platelet count<90×10^9/L; hemoglobin below the lower limit of normal; serum creatine kinase (CK) >3×ULN; blood phosphorus <0.8 mmol/L; serum creatinine (SCr) > 1×ULN.
* Diabetes mellitus or Poorly controlled Thyroid Diseases.
* Poorly controlled hypertension (systolic blood pressure> 140mmHg, or diastolic blood pressure> 90 mmHg) with hypertension -related retinal lesions.
* Immunodeficiency or autoimmune diseases including but not limited to inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, scleroderma, Sjogren's syndrome, autoimmune thrombocytopenia, etc.
* Psychiatric and nervous system disorders, including history of psychiatric illness or with family history (especially depression, depressive tendencies, epilepsy and hysteria, etc.)
* Severe cardiovascular diseases (New York Heart Association functional class (NYHA) Ⅲ level and above, myocardial infarction occurred within past 6 months or PTCA performed within past 6 months, unstable angina, uncontrolled arrhythmias).
* Serious blood disorders (all kinds of anemia, hemophilia, etc.)
* Severe kidney disease (chronic kidney disease, renal insufficiency, etc.)
* Serious digestive diseases (gastrointestinal ulcers, colitis, etc.)
* Severe respiratory disease (pneumonia, chronic obstructive pulmonary disease, interstitial lung disease, etc.)
* Retinal disease (retinal exfoliation, macular hole, retinal tumors, etc.)
* Malignancies.
* Function organs transplant.
* Allergies or severe allergies, especially allergic to study drugs or any ingredients of the study drugs.
* Evidence of alcohol or drug abuse (average alcohol consumption male> 40g / day, female> 20g / day).
* Women who are pregnant or lactating or to be pregnant during the study period.
* Participated in other clinical trials 3 months prior to the screening.
* Unwilling to sign the informed consent and adhere to treatment requirements.
* Other conditions not suitable for study judged by investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBsAg negative. | 72 weeks
  Percentage of Participants with HBsAg <0.05 IU/mL

CONTACTS AND LOCATIONS:
Locations (34):
- China (34):
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Peking university Peoole's hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The second xiangya hospital of central south university, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - The Peoole's hospital of Chizhou, Chizhou
  - The First Affiliated Hospital of Army Medical University, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Mengchao hepatobiliary hospital of Fujian medical university, Fuzhou
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Heze Municipal Hospital, Heze
  - Shandong Public Health Clinical Center, Jinan
  - Hebei petro china central hospital, Langfang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Hospital of Nanjing, Nanjing
  - Pingxiang NO.2 People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - The Peoole's hospital of Qingyuan, Qingyuan
  - The Sixth People's Hospital of Shenyang, Shenyang
  - Shijiazhuang Hospital of Traditional Chinese Medicine, Shijiazhuang
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - The Second People's Hospital of Tianjin, Tianjin
  - Tianjin Third Central Hospital, Tianjin
  - Tongji medical college of Hust, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an
  - The third affiliated hospital of Xingxiang medical university, Xingxiang
  - Yanbian University Hospital, Yanbian
  - Henan People's Hospital, Zhengzhou
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou

IPD SHARING:
Plan to Share IPD: No